CLINICAL TRIAL: NCT01173003
Title: An Open Label Study of 400 mcg Sublingual Misoprostol Following Mifepristone 200 mg for Abortion up to 63 Days LMP
Brief Title: Expansion Study of a Simplified Regimen of Medical Abortion Thru 63 Last Menstrual Period (LMP) in Tunisia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: Centre de Formation et de la Recherche, Tunisia (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1.1.7
Record Dates: First submitted 2010-07-28; First posted 2010-07-30 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Induced Abortion
Keywords: Medical abortion; mifepristone; misoprostol; Tunisia
MeSH Terms: interventions — Mifepristone; Misoprostol

INTERVENTIONS:
Drug: Mifepristone, misoprostol

SUMMARY:
This open-label study is being conducted to determine whether national expansion of a 400 mcg of sublingual misoprostol (i.e., under the tongue) taken 24 hours following administration of mifepristone 200 mg is effective and acceptable to new abortion providers in 14 regions.

The goal of this study is to provide answers to the following four questions:

1. What is the effectiveness of this regimen of medical abortion with mifepristone followed by 400 mcg sublingual misoprostol up to 63 days since the last menstrual period (LMP)?
2. Are the side effects with sublingual use tolerable for women?
3. Is sublingual administration of misoprostol acceptable to women?
4. Are women satisfied with counseling and services received in new centers offering medical abortion?

ELIGIBILITY:
Inclusion Criteria:

* Women presenting for medical abortion who consent to participate
* Possibility of final gestational age of less than or equal to 63 days
* General good health
* Willing to provide contact information for purposes of follow-up

Exclusion Criteria:

* Conditions which contraindicate the use of mifepristone or misoprostol
* Women presenting for medical abortion who do not consent to participate

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 688 (Actual)
Dates: Start 2009-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Need for surgical completion for incomplete abortions or ongoing viable pregnancies at follow up visit Study day 15. | 2 weeks after mifepristone administration

SECONDARY OUTCOMES:
Side effects | 48 hours
Acceptability for women | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, MD, MPH, Study Chair — Gynuity Health Projects; Rasha Dabash, MPH, Study Director — Gynuity Health Projects; Selma Hajri, MD, Principal Investigator — Reproductive Health Consultant; Mongia Ben Attia, MD, Principal Investigator — Office Nationale de la Famille et de la Population; N Gueddana, MD, Study Chair — ONFP; Fatma Temimi, MD, Principal Investigator — ONFP; E Hassairi, Principal Investigator — ONFP
Locations (1):
- Centres (14) de Planification Familiale de L'ONFP, Tunis, Various, Tunisia